CLINICAL TRIAL: NCT00169663
Title: Brushite Stones: A Registry and Database of Clinical and Laboratory Findings
Brief Title: Brushite Kidney Stones: A Registry and Database of Clinical and Laboratory Findings
Status: Completed | Type: Observational
Sponsor: Indiana Kidney Stone Institute (Other)
Responsible Party: James Lingeman, MD, IU Health Physicians Urology
Other Study IDs: 03-049
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Nephrolithiasis
Keywords: Brushite Kidney Stones; Nephrolithiasis
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Brushite kidney stones are a unique form of calcium phosphate stones that have a tendency to recur quickly if patients are not aggressively treated with stone prevention measures. Little research has been undertaken to better understand the clinical history and potential urinary abnormalities that may predispose one to these troublesome kidney stones.

DETAILED DESCRIPTION:
Multiple treatment options are available for the treatment of kidney or ureteral calculi. Treatment options include shock wave lithotripsy (SWL; shock waves are transmitted through the body wall and focused onto the stone to break the stone into gravel), percutaneous nephrolithotomy (PNL; a small flank incision is made and a telescope inserted into the kidney to allow stone fragmentation and removal from the patient), and ureteroscopic lithotripsy (URS; a small telescope is inserted into the ureter or kidney and a laser is used to break up the stone into gravel).

Brushite is a unique form of calcium phosphate kidney stone that often has sub-optimal stone fragmentation with shock wave lithotripsy (Heimbach et al, 1999). Due to its SWL resistance, brushite patients often undergo more invasive treatments such as URS or PNL to achieve a stone free status. Brushite patients often have multiple stones and have a high likelihood of developing recurrences (new stone formation or regrowth of existing stone fragments), often within the first year after surgery. These patients may also have a history of anatomical abnormalities of the urinary tract or a history of prior renal or ureteral surgery (Klee et al, 1991).

A thorough review of the clinical, radiological and metabolic data of brushite patients has the potential to clarify a number of important points. Many patients with brushite stones often have a history of non-brushite stones (e.g. calcium oxalate) predating the development of brushite stones and historical review is needed to define the factors contributing to this shift in stone composition. In addition, it has been shown that CT attenuation values can be used to predict stone composition (Joseph et al, 2002). As a result, it is crucial to review the radiologic appearance of known brushite stones to identify specific radiographic characteristics and possibly allow a radiographic diagnosis of brushite to be established. Finally, very little information has been reported on the urinary abnormalities in brushite patients. By carefully examining 24 hour urine data in a large population of brushite patients, information may be identified that can be used to provide improved management of specific abnormalities to prevent stone recurrences.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients of Methodist Urology in Indianapolis, IN over the age of 18 with brushite stones.

Exclusion Criteria:

1. Patients unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of Methodist Urology in Indianapolis, IN who have a stone analysis of 100% brushite stone
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2003-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To review the clinical and laboratory findings in a population of brushite patients who have been treated at Methodist Urology, LLC | one year

CONTACTS AND LOCATIONS:
Overall Officials: James E Lingeman, MD, Principal Investigator — IU Health Physicians Urology
Locations (1):
- Methodist Hospital, Indianapolis, Indiana, United States